CLINICAL TRIAL: NCT06015672
Title: Duke Accelerated Transcranial Magnetic Stimulation for Focal Hand Dystonia
Brief Title: Accelerated TMS for Focal Hand Dystonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00112239
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Isolated Focal Hand Dystonia
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double-arm crossover study design with subjects receiving TMS at two different intensities
Who Masked: Participant, Outcomes Assessor
Masking Description: The TMS intensity delivered at each TMS visit will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TMS to primary somatosensory cortex (Active Comparator): Participants received TMS sessions at primary somatosensory cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS at low amplitude to primary somatosensory cortex (Sham Comparator): Participants receive TMS at a cortical target at smaller amplitude
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Participants will have two accelerated transcranial magnetic stimulation (TMS) visits. Each TMS visit will be separated by 5 months. During each TMS visit, they will receive four TMS sessions, each separated by 60 minutes of rest.

SUMMARY:
This study aims to investigate the impact of accelerated transcranial magnetic stimulation (TMS) on brain function and behavior in patients with focal hand dystonia. Previous research demonstrated that individualized TMS improved dystonic behavior after one session. Building on this, the current study administers four TMS sessions in a day, with assessments conducted in four weeks, twelve weeks, and 20 weeks after each session. The research involves 8 in-person and 6 virtual visits focused on functional MRI brain scans and writing behavior analysis. The potential risk of seizures from TMS is mitigated through careful screening, adhering to safety guidelines. The study's main benefit is enhancing dystonic behavior and deepening the understanding of brain changes caused by TMS in focal hand dystonia, paving the way for further advancements in clinical therapy for this condition.

DETAILED DESCRIPTION:
The primary aim of this research is to investigate the impact of transcranial magnetic stimulation (TMS) on both brain function and behavioral outcomes among individuals suffering from focal hand dystonia. A preliminary examination of a previous TMS study carried out by our team revealed that the application of TMS, using personalized, fMRI-guided brain targeting and interleaved TMS delivery during motor tasks, has the potential to modify brain activity and ameliorate dystonic behavior after a single session of TMS in patients with focal hand dystonia. This present study seeks to build upon these promising findings by administering four TMS sessions in a single day, interspersed with four rest intervals, a protocol referred to as "accelerated TMS." The investigation will consist of a total of eight in-person appointments. Participants with focal hand dystonia will receive accelerated TMS during two in-person visits. Following each TMS session, participants will evaluate changes in brain function and behavior. During the assessment visits, individuals will undergo functional MRI brain scans and engage in writing tasks on an electronic tablet. The principal risk associated with TMS is the possibility of inducing a seizure. However, this study will strictly adhere to safety guidelines, utilizing TMS levels that have not previously been linked to seizures in properly screened individuals. Notably, the dosages of TMS proposed for use in this study have not caused seizures in healthy volunteers. To further mitigate the risk of seizures, potential subjects will undergo medical screening for any known factors that could predispose them to seizures. The primary advantage of this study lies in its potential to enhance dystonic behavior in patients with focal hand dystonia, while also deepening our comprehension of the foundational changes in brain function before and after TMS intervention for focal hand dystonia. The discoveries stemming from this investigation will pave the way for future research endeavors aimed at advancing brain stimulation as a viable clinical therapy for focal hand dystonia.

ELIGIBILITY:
Inclusion Criteria:

* 18yrs and older
* Diagnosed with isolated focal hand by Neurologist
* Right-hand dominant
* Must be able to sign an informed consent
* Must be literate

Exclusion Criteria:

* Other neurological movement disorders diagnoses including other types of dystonia, Parkinsonism, or essential tremor
* History of seizure disorder
* Concomitant medications are known to decrease seizure threshold
* Illicit drug use
* No TMS therapy for another indication within one month of this research study
* Botulinum toxin injections within 3months of the research study
* Medications used for symptom treatment of dystonia including anticholinergic, benzodiazepines, and muscle relaxants among others within one month of the study
* No physical or occupational therapy of the hand within one month of the study
* Any contraindications to MRI or TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in behavioral writing measure | Baseline, 4 weeks, 12 weeks, 20 weeks, 24, weeks, 32 weeks and 40 weeks
  Using change in peak accelerations to assess writing behavior
Change in brain connectivity in the motor network | Baseline, 12 weeks, 20 weeks and 32 weeks
  Using functional magnetic resonance imaging of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Bukhari-Parlakturk, MD PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noreen Bukhari-Parlakturk, Patrick Mulcahey, Michael Lutz, Rabia Ghazi, Ziping Huang, Moritz Dannhauer, Zeynep Simsek, Skylar Groves, Mikaela Lipp, Michael Fei, Tiffany Tran, Eleanor Wood, Lysianne Beynel, Burton Scott, Pichet Termsarasab, Chris Petty, Hussein R Al-Khalidi, James Voyvodic, Lawrence G. Appelbaum, Simon Davis, Andrew Michael, Angel Peterchev, Nicole Calakos. "Functional MRI-guided individualized TMS modifies motor network and reduces writing dysfluency in Focal Hand Dystonia." Human Brain Mapping Conference. Montreal, Canada. July 22-26, 2023. virtual poster presentation.
- [Background] Noreen Bukhari-Parlakturk, Patrick Mulcahey, Michael Lutz, Rabia Ghazi, Ziping Huang, Moritz Dannhauer, Zeynep Simsek, Skylar Groves, Mikaela Lipp, Michael Fei, Tiffany Tran, Eleanor Wood, Lysianne Beynel, Burton Scott, Pichet Termsarasab, Chris Petty, Hussein R Al-Khalidi, James Voyvodic, Lawrence G. Appelbaum, Simon Davis, Andrew Michael, Angel Peterchev, Nicole Calakos. "Functional MRI-guided individualized TMS modifies motor network and reduces writing dysfluency in Focal Hand Dystonia." Samuel Belzberg 6th International Dystonia Symposium. Dublin, Ireland. June 1-3, 2023. poster presentation.
- [Background] Bukhari-Parlakturk N, Lutz MW, Al-Khalidi HR, Unnithan S, Wang JE, Scott B, Termsarasab P, Appelbaum LG, Calakos N. Suitability of Automated Writing Measures for Clinical Trial Outcome in Writer's Cramp. Mov Disord. 2023 Jan;38(1):123-132. doi: 10.1002/mds.29237. Epub 2022 Oct 13. PMID 36226903
- [Background] Dannhauer M, Huang Z, Beynel L, Wood E, Bukhari-Parlakturk N, Peterchev AV. TAP: targeting and analysis pipeline for optimization and verification of coil placement in transcranial magnetic stimulation. J Neural Eng. 2022 Apr 21;19(2):10.1088/1741-2552/ac63a4. doi: 10.1088/1741-2552/ac63a4. PMID 35377345